CLINICAL TRIAL: NCT06836518
Title: Serum Sialic Acid as a Novel Biomarker in the Diagnosis of Hepatocellular Carcinoma
Brief Title: Sialic Acid in Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eman Khalifa Elsayed, Assistant Lecturer of Tropical Medicine and Gastroenterology, Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med-25-2-1MD
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy persons: The study group will include normal healthy persons who will be selected randomly.
  Interventions: Diagnostic Test: serum sialic acid
- cirrhotic patients: The study group will include patients diagnosed with liver cirrhosis with no detected hepatic focal lesion by ultrasound.
  Interventions: Diagnostic Test: serum sialic acid
- cirrhotic patients with hepatocellular carcinoma: The study group will include patients with liver cirrhosis and hepatocellular carcinoma. All causes of liver cirrhosis will be accepted. HCC will be assessed by triphasic CT or MRI.
  Interventions: Diagnostic Test: serum sialic acid

INTERVENTIONS:
Diagnostic Test: serum sialic acid — measurement of serum sialic acid to evaluate its efficacy in the diagnosis of hepatocellular carcinoma

SUMMARY:
Hepatocellular carcinoma (HCC) accounts for approximately 90% of the cases of liver cancer and is associated with high morbidity and mortality.

The increased sialic acids(SAs) in tumor cells are mainly caused by the special metabolic flux and aberrant expression of sialyltransferases/sialidases, The high sensitivity of sialic acids in or plasma as a tumor marker has been reported in various cancerous conditions the level of sialic acid(SA) activity was found to offer highly specific and sensitive tumor biomarker for diagnosis and follow up of HCC post-therapy.

DETAILED DESCRIPTION:
Liver cancer is a growing global health challenge, with an estimated annual incidence of >1 million cases worldwide by 2025.

Hepatocellular carcinoma (HCC) accounts for approximately 90% of the cases of liver cancer and is associated with high morbidity and mortality.

The most prominent risk factors for HCC include hepatitis B (HBV), hepatitis C (HCV) viral infections and non-alcoholic steatohepatitis (NASH), which can lead to liver fibrosis and cirrhosis.

Other risk factors include heavy alcohol consumption, non-alcoholic fatty liver disease (NAFLD), consumption of aflatoxins, obesity associated with metabolic syndrome, type 2 diabetes (T2D), and tobacco smoking.

Sialic acids (SAs) are a subset of nine carbon acidic sugars that contain approximately fifty derivatives of neuraminic acids. The most common sialic acid derivatives found in mammals are N-acetylneuraminic acid (Neu5Ac) and N-glycolylneuraminic acid (Neu5Gc).

Sialic acid (SA) structural diversity leads to many biological functions, including antiviral activity, antioxidant activity, anti-adhesion activity , anti-inflammatory property, and improving learning and memory, promoting bone growth and prebiotics .

SA can participate in important pathological and physiological processes and can be used as nutrition, drugs and drug carriers to prevent diseases. Therefore, SA is a promising active substance, which can improve human health.

SAs on tumor cell surfaces are aberrantly expressed during tumor transformation and malignant progression. In general, hypersialylation is frequently observed in tumor tissues compared to corresponding normal tissue.

The increased SAs in tumor cells are mainly caused by the special metabolic flux and aberrant expression of sialyltransferases/sialidases.

Abnormal expression of SA is atypical symbol of tumor cells. β-galactoside α2,6 sialyl transferases is closely related to tumorigenesis and tumor progression. High levels of β-galactoside α2,6-sialyltransferases mediated tumorigenesis and metastasis in HCC cells by activating the Wnt/β-catenin pathway.

The high sensitivity of SAs in serum or plasma as a tumor marker has been reported in various cancerous conditions. Quantification of total SAs or glycolipid-bound sialic acids in serum is helpful to improve the accuracy of clinical diagnoses and therapies.

The level of SA activity was found to offer highly specific and sensitive tumor biomarker for HCC diagnosis and follow up of HCC post-therapy.

ELIGIBILITY:
Inclusion Criteria:

* The study will include normal persons, patients with liver cirrhosis and HCC patients attending to the outpatient clinic or inpatient section of the department of Tropical medicine and Gastroenterology and Radiological department at Sohag University Hospital will be included.

Exclusion Criteria:

* 1- Patients aged < 18 or > 70 years. 2- Patients with other malignancy rather than HCC. 3- Patients with history of prior intervention or systemic chemotherapy for HCC.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include normal persons, patients with liver cirrhosis and HCC patients attending to the outpatient clinic or inpatient section of the department of Tropical medicine and Gastroenterology and Radiological department at Sohag University Hospital will be included.
  HCC will be assessed by ultrasonography, alpha fetoprotein plus triphasic CT or MRI.
  Group I:
  The study group will include normal healthy persons who will be selected randomly.
  Group II:
  The study group will include patients diagnosed with liver cirrhosis with no detected hepatic focal lesion by ultrasound.
  Cirrhosis will be determined according to clinical, serological and radiological findings.
  Group III:
  The study group will include patients with liver cirrhosis and HCC. All causes of liver cirrhosis will be accepted. HCC will be assessed by triphasic CT or MRI.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Serum Sialic Acid | one year
  measurement of serum sialic acid concentration according to ELISA method to evaluate its diagnostic efficacy in hepatocellular carcinoma

IPD SHARING:
Plan to Share IPD: Undecided